CLINICAL TRIAL: NCT02114749
Title: Development of Tools for Respiration and Circulation Studies and Exploration, Their Mutual Interactions and the Functions Involved in the Daily Life in Healthy Volunteers
Brief Title: Development of Tools for Respiration and Circulation Exploration
Acronym: MAPO-RCVQ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Université Joseph Fourier (Other); Centre National de la Recherche Scientifique, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: University Hospital, Grenoble
Record Dates: First submitted 2014-03-14; First posted 2014-04-15 (Estimated); Last update posted 2018-05-18 (Actual); Status verified 2018-05

CONDITIONS: Motor Activity
Keywords: Healthy volunteers; Physiological variables : respiration and circulation
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- volunteers in daily life activities (Experimental): a set of wearable respiration and cardiac monitoring devices
  Interventions: Device: a set of wearable respiration and cardiac monitoring devices

INTERVENTIONS:
Device: a set of wearable respiration and cardiac monitoring devices — feasibility of methods for detecting physiological state changes from a set of wearable respiration and cardiac monitoring devices
  Other Names: Equivital® from Hidalgo Ltd UK,; VISURESP from RBI Instrumentation France,; Finometer® from Finapres Medical Systems NL

SUMMARY:
This study is aimed to develop analysis methods and measurements tools for physiological variables : respiration, circulation and their mutual interactions and with the functions involved in the daily life in healthy volunteers (drinking, eating, sleeping, coughing...). The devices that are used are non invasive. The development of these tools needs to be validated on physiological signals obtained in healthy volunteers.

DETAILED DESCRIPTION:
The analysis and interpretation of a record consist, for example, to measure the amplitude of the respiratory modulation of the cardiac period, a witness of the level of the subject's sympathetic activity.

To do this, a mathematical model of this oscillation is adjusted on the experimental data, and its characteristics (amplitude, phase, non-linearity...) are considered indexes of the interaction to be compared with the same characteristics in other conditions.

The transition to clinical applications requires validation of the developed tools on physiological signals recorded on healthy volunteers in a non-clinical environment, avoiding extra psychological stress in the Protocol followed.

Whether it is for the development of tools or their validation, it is essential that the sensors used are non-invasive.

Recorded situations are those of everyday life, such as working (only sedentary work are envisaged), eat, talk, rest and move from one place of life to another one.

ELIGIBILITY:
Inclusion Criteria:

* healthy, major and socially insured human subjects

Exclusion Criteria:

* deprived of liberty, hospitalized and protected human subjects

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-02-24 (Actual); Primary Completion 2017-12-13 (Actual); Study Completion 2017-12-13 (Actual)

PRIMARY OUTCOMES:
Feasibility and use of developed methods and tools in clinical or fundamental research protocols or in systems for physiological monitoring in humans | up to 24 months
  The new tools for identification and monitoring of the physiological state of a subject will be developed from a set of non-invasive measures at rest. Resulting physiological state identification will then be validated on registrations on the same subjects in different daily life circumstances.

CONTACTS AND LOCATIONS:
Overall Officials: Briot Raphaël, MD, Principal Investigator — University Hospital, Grenoble
Locations (2):
- France (2):
  - TIMC - pavillon Taillefer - CHU, Grenoble
  - University Hospital, Grenoble

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fiamma MN, Straus C, Thibault S, Wysocki M, Baconnier P, Similowski T. Effects of hypercapnia and hypocapnia on ventilatory variability and the chaotic dynamics of ventilatory flow in humans. Am J Physiol Regul Integr Comp Physiol. 2007 May;292(5):R1985-93. doi: 10.1152/ajpregu.00792.2006. Epub 2007 Jan 11. PMID 17218438
- [Background] Ben Lamine S, Calabrese P, Perrault H, Dinh TP, Eberhard A, Benchetrit G. Individual differences in respiratory sinus arrhythmia. Am J Physiol Heart Circ Physiol. 2004 Jun;286(6):H2305-12. doi: 10.1152/ajpheart.00655.2003. Epub 2004 Jan 29. PMID 14751864
- [Background] Eberhard A, Calabrese P, Baconnier P, Benchetrit G. Comparison between the respiratory inductance plethysmography signal derivative and the airflow signal. Adv Exp Med Biol. 2001;499:489-94. doi: 10.1007/978-1-4615-1375-9_79. No abstract available. PMID 11729931
- [Background] Emeriaud G, Eberhard A, Benchetrit G, Debillon T, Baconnier P. Calibration of respiratory inductance plethysmograph in preterm infants with different respiratory conditions. Pediatr Pulmonol. 2008 Nov;43(11):1135-1141. doi: 10.1002/ppul.20923. PMID 18846561
- [Background] Fontecave-Jallon, Gumery P-Y, Calabrese P, Briot R, Baconnier P. A wearable technology revisited for cardio-respiratory functional exploration : Stroke volume estimation form respiratory inductive plethysmography. International journal of eHealth and Medical Communications, 4, 2013
- See also: web site laboratory Techniques de l'Ingénierie Médicale et de la Complexité - Informatique, Mathématiques et Applications, Grenoble (TIMC-IMAG) — http://www-timc.imag.fr/